CLINICAL TRIAL: NCT06800222
Title: The Effectiveness of Modern Physical Agents in Treating Pelvic Floor Dysfunctions, Improving Functional State, Life Quality, and Biosocial Functions During First-stage Pelvic Rehabilitation.
Brief Title: Effectiveness of Modern Physical Agents in the Treatment of Pelvic Floor Dysfunctions
Acronym: EMPHAT-PFD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Venta Donec, Physical medicine and rehabilitation physichian, Phd, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-02 V-3
Record Dates: First submitted 2024-10-26; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Pelvic Floor Dysfunctions
Keywords: pelvic floor dysfunctions; pelvic pain; urgency; incontinece; vaginismus; constipation; erectile dysfunction; irritable bladder
MeSH Terms: conditions — Pelvic Pain; Vaginismus; Constipation; Erectile Dysfunction; Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Subjects will receive classical rehabilitation interventions together with modern physical agents
  Interventions: Other: modern agents rehab
- Control (Other): subject will receive only classical rehabilitation interventions
  Interventions: Other: classical rehab

INTERVENTIONS:
Other: modern agents rehab — rehabilitation interventions containing modern physical agents together with classical interventions
  Arms: Intervention group
Other: classical rehab — classical rehabilitation interventions
  Arms: Control

SUMMARY:
This clinical trial aims to determine whether adding modern physical agents (high-intensity laser therapy, magnetotherapy, radial shock wave therapy, kinesiotaping) in conjunction with classical rehabilitation interventions produces superior outcomes in treating pelvic floor dysfunction compared to classical rehabilitation interventions alone. It will also assess the safety of these agents in the context of pelvic floor dysfunction rehabilitation. The main questions it aims to answer are:

Does adding modern physical agents to the treatment of pelvic floor dysfunction improve symptoms, impairments in functional state, quality of life, and biosocial functions more effectively than classical interventions alone?

Participants who experience pelvic floor dysfunction during primary rehabilitation will receive:

Either an individualized rehabilitation intervention plan comprising 20 classical procedures in combination with modern physical agents or classical interventions alone. Rehabilitation will take place in the outpatient rehabilitation department. Patients will visit the clinic for a comprehensive functional state assessment and then for individualized procedures; the entire plan will be delivered over three months, after which participants will return for follow-up checkups and assessments after the procedures and again after six months.

DETAILED DESCRIPTION:
After subjects are included in the research, two groups (interventional-modern agents rehab and control-classical rehab) of 125 patients each will be formed through concealed randomization. A person not connected with the study will use a random number generator to allocate subjects to the groups.

The rehabilitation process for all subjects will include a comprehensive functional assessment, setting short-term and long-term individualized goals for each subject, prescribing and implementing a primary outpatient rehabilitation plan involving various rehabilitative interventions. Once the plan is implemented, the physical medicine and rehabilitation (PMR) physician will thoroughly assess the rehabilitation results. An observation period will follow, during which learned self-help techniques will be integrated into daily life. After six months, all subjects will be reassessed by a PMR physician.

Process:

After inclusion, all participants will be thoroughly assessed by a qualified PMR physician specializing in pelvic floor dysfunction rehabilitation. Following all functional assessments, an individualized primary outpatient rehabilitation plan will be agreed upon with the patient, comprising 20 rehabilitative interventions. Depending on the group to which the subject is randomized, the individualized rehabilitation interventions will either consist of classical interventions (such as physiotherapy, occupational therapy, electrical stimulation, etc.) for the control group, or classical interventions combined with modern physical agents for the interventional group.

During the rehabilitation period, the rehabilitation team will monitor subjects in both groups for any side effects from the rehabilitation interventions. Subjects will also have the option to inform and consult a PMR physician as often as needed in case of side effects or intolerance to prescribed interventions.

The PMR physician will conduct thorough functional assessments again after rehabilitation and after six months.

Methods to assess functioning and pelvic floor dysfunctions:

Before rehabilitation:

Detailed questioning regarding the history of pelvic floor dysfunction, other treatments received, general health, and relevant psychosocial factors will precede setting an individualized rehabilitation plan for pelvic floor dysfunctions. The four-item patient health questionnaire for anxiety and depression ( PHQ-4 ) will be used when indicated. Subjects may be asked to fill out a 3-day bladder diary, a diary on bowel incontinence events, a male patients' diary on erection/ejaculation quality and satisfaction with sexual activity, or a pain questionnaire covering pain diagrams and intensity assessments, questions on pain quality, duration, and exacerbation/or alleviation factors, and changes over time.

A trained PMR physician will conduct a thorough clinical examination (including posture, perineum, and digital external and internal pelvic floor muscle assessment) and, when possible, functional testing of slow and quick muscle fibers endurance.

Functional assessment of the abdominal wall (for diastasis, abdominal muscle activity during a curl-up task, straight leg raise task) and pelvic floor muscle morphological and functional evaluation will be performed using two and three-dimensional (2D/3D) ultrasound (transabdominal and transperineal).

After rehabilitation:

To assess subjective experiences and attitudes towards received outpatient rehabilitation, all subjects will complete a self-reported questionnaire about symptom improvement based on global improvement rating scales. The questionnaire will also contain open-ended questions about patient expectations, experiences with learned self-help techniques, attitudes, and suggestions for the rehabilitation team regarding pelvic floor dysfunction rehabilitation. Subjects will rate the perceived helpfulness of each received rehabilitative intervention on a numeric 0-10 scale (where 0 is 'not helpful at all' and 10 is 'maximally helpful').

A thorough clinical examination (including perineum, digital external and internal pelvic floor muscle assessment) and, when possible, functional testing of slow and quick muscle fibers endurance will be conducted by a trained PMR physician.

Functional assessment of the abdominal wall (for diastasis), abdominal muscles, and pelvic floor muscle morphological and functional evaluation will be performed using 2D/3D ultrasound (transabdominal and transperineal).

When indicated (depending on symptoms and dysfunctions), subjects may be asked to fill out a 3-day bladder diary, a pain questionnaire, or diaries on bowel incontinence events and male sexual function.

The PHQ-4 will be used.

After six months:

detailed questionnaire on changes in pelvic floor dysfunction symptoms post-rehabilitation, other treatments received, general health, and other psychosocial factors will be conducted by a PMR physician to determine if further rehabilitation interventions are necessary. When indicated, subjects may be asked to fill out a 3-day bladder diary, a pain questionnaire, or other condition-specific diaries.

The PHQ-4 will be used for all subjects. A thorough clinical examination (including perineum, digital external and internal pelvic floor muscle assessment) and, when possible, functional testing of slow and quick muscle fibers endurance will be conducted by a trained PMR physician.

Functional assessment of the abdominal wall (for diastasis), abdominal muscles, and pelvic floor muscle

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years old.
2. One or more signs characteristic of pelvic floor dysfunctions are identified: elimination function disorders, pelvic organ prolapse, scar(s) (and lack of tissue mobility) in the perineum, pelvic floor muscle tone/strength disorders (hypoactivity/hyperactivity), neuromuscular control disorders, sexual dysfunctions, pain in the pelvis, perineum.
3. Not a single exclusion criterion has been established.
4. Subjects capable of signing informed consent.

Exclusion Criteria:

1. Oncological diseases or being actively investigated for oncological diseases.
2. Any contraindications to methods of functional state examination or physical agents in the pelvic area that will be used in the study
3. Individuals who refuse a detailed clinical examination of the perineum and pelvic floor muscles, functional testing, and/or functional ultrasound examination.
4. Patients with urinary tract, prostate, genital, and other infections.
5. Patients with inflammatory bowel diseases (ulcerative colitis, Crohn's disease, etc.).
6. Persons for whom other health care professionals have already planned treatment of pelvic dysfunctions or other diseases during the expected participation period in the study that may interfere with participation in the study and/or significantly change the health status of the patient's pelvic floor.
7. Pregnant or planning to become pregnant during the expected period of rehabilitation interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-09-09 (Estimated); Study Completion 2029-09-09 (Estimated)

PRIMARY OUTCOMES:
Overall change in bothering pelvic floor symptoms according to Global Rating of Change (GRC) scales | 3 months
  After rehabilitation, the overall change in bothering pelvic floor dysfunction symptoms according to Global Rating of Change (GRC) scales will be assessed.
  The Global Rating of Change (GRC) Scale is a tool used to assess a patient's perceived change in health status over time. The minimum value is 0, indicating "no change." The maximum value is 10, indicating "a very great deal better." Higher scores on the GRC Scale reflect a better outcome, showing greater perceived improvement in the patient's symptoms.

SECONDARY OUTCOMES:
Overall change in urinary dysfunction symptoms | 3 months and 6 months
  The overall change in urgency and incontinence symptoms (if applicable) will be assessed by 3-day bladder dairy after rehabilitation and at the follow-up.
  A 3-day bladder diary is when, over three days, patients record details about their urinary habits, including the frequency and volume of urination, fluid intake, and any incontinence episodes. This diary helps healthcare providers assess lower urinary tract symptoms and develop appropriate treatment plans. Additionally, in this study, diary data will help to monitor changes in minimal/maximum volume, average volume during urination, incontinence severity, and changes in incontinence episodes.
Overall change in fecal incontinence | 3 months and 6 months
  A diary of accidents will assess the overall change in fecal incontinence (if applicable).
  Subjects will be asked to record each incontinence event and provide information about the frequency, timing, and possible triggers of incontinence episodes. This detailed record helps healthcare providers identify patterns, understand the severity of the condition, and develop personalized treatment plan to improve the quality of life. In this study, the diary will help to assess the overall change in fecal incontinence symptoms, frequency, and severity.
Overall change in pelvic pain | 3 months and 6 months
  The overall change in pelvic pain (if applicable) will be assessed using a questionnaire with the following questions: 1) Pain intensity at different times and during various activities, such as day/night, walking, changing body positions, lying/sitting/standing, during sexual activity, urination, and defecation, as well as after sexual activity, urination, and defecation. This will be measured by the Numeric Pain Rating Scale (NPRS), where 0 indicates "no pain at all," and 10 indicates "worst imaginable pain." 2) Pain duration during the day/night, while walking, changing body positions, and while lying/sitting/standing, with possible answer choices: Constant (always the same intensity); Constant (pain intensity varies); Often felt (pain-free periods shorter than 6 hours); Intermittent; I did not feel pain.
  3) Pain localization will be assessed using a pain diagram, allowing subjects to indicate where they experience pain by marking specific areas.
Overall change in male sexual function | 3 months and 6 months
  If applicable, changes in male sexual function will be assessed through a self-evaluation diary that subjects experiencing sexual dysfunction will be asked to fill out during participation. In this diary, subjects will need to self-report events of sexual activity (intercourse or masturbation), its duration, the dominant body position, the quality of erection during sexual activity as a percentage, where 0% indicates no erection at all (flaccid penis), 50% erection is sufficient for vaginal penetration, and 100% erection is a maximally hard penis (maximum erection). They will also evaluate the quality of ejaculation during sexual activity with possible options: failed to ejaculate, premature ejaculation, delayed ejaculation, or good (normal, timely) ejaculation. Subjects will report overall pleasure achieved with the activity on a scale from 0-100% (0 indicating no satisfaction at all, 100% indicating maximal satisfaction/pleasure).
Change in pelvic floor muscle contraction: ability to contract and relax pelvic floor muscles | 3 months and 6 months
  ability to contract and relax pelvic floor muscles (voluntary and non-voluntary) will be assessed clinicaly through inspection and palpation following the recomendations of International Continence Society for pelvic floor clinical assessment. Additionally voluntary and non-voluntry contraction/relaxation will be assessed through functional ultrasound (visualizing the contractions and relaxation) as well as measuring the changes in levator ani anteriorposterior line distance during efforts to provoke voluntary and non-voluntary (cough test/straining) contraction and relaxation. The Levator ani anterior-posterior distance with ultrasound will be measured transperinealy from a defined anterior point (the pubic symphysis) to a posterior point (the anorectal junction), measured in milimeters.
Change in pelvic floor painfulness from palpation | 3 months and 6 months
  During clinical palpation of the pelvic floor, subjects will be asked to indicate if they feel any pain and to specify its intensity on the Numeric Pain Rating Scale (NPRS) (0 = no pain at all, 10 = worst imaginable pain). The anatomical areas where tissues are painful to palpation and the pain intensity will be documented in the assessment protocol.
Change in pelvic floor muscle endurance | 3 months and 6 months
  If applicable, pelvic floor muscle endurance will be assessed through clinical examination as suggested by the International Continence Society. Endurance is expressed as the length of time, up to 10 seconds, that maximal voluntary contractions of the pelvic floor muscles can be sustained before strength is reduced by 35% or more. The number of repetitions (up to 10) of maximal voluntary contractions will then be recorded, allowing four seconds of rest between each contraction. After a one-minute rest, the number (up to 15) of one-second maximal voluntary contractions will be assessed.
Change in pelvic floor muscle strenght | 3 months and 6 months
  Pelvic floor muscle strength will be assessed clinically by a modified Oxford scale. (MOS). The MOS is used to rate pelvic floor muscle contractility on a scale of 0-5: 0, no contraction; 1, minor muscle 'flicker'; 2, weak muscle contraction without a circular contraction; 3, moderate muscle contraction; 4, good muscle contraction; and 5, strong muscle contraction against resistance by the examining finger. Additionally (if applicable), women will undergo 3D transperineal functional ultrasound testing. The reduction in hiatal area (in square mm) and anteroposterior diameter (mm) during maximal induced pelvic ﬂoor muscle contraction will be measured, and the percentage change will be identified. The formula for counting the change will be: difference = ((Measurement at rest - Measurement at squeeze/straining )/Measurement at rest ) × 100%. If signs of levator ani avulsion or hiatal ballooning, asymmetry in contraction is notified, this will be noted in the assessment protocol.
Change in diastasis recti | 3 months and 6 months
  If applicable (in cases of diastasis recti), the inter-rectus distance (IRD) change after rehabilitation and at the 6-month follow-up will be measured with transabdominal ultrasound at four locations, with the subject lying on their back in a resting position: AU1: ½ of the superior umbilical border-xiphoid distance; AU2: ¼ of the superior umbilical border-xiphoid distance; U: the superior umbilical border; BU: ¼ of the superior umbilical border-pubis distance. The change in percentage from the measured values before rehabilitation will be calculated using the formula: ((IRD in mm {baseline measurement} - IRD in mm{following measurement}) / IRD in mm {baseline measurement} * 100%). The ultrasound diagnostic criteria we will use for diagnosing diastasis recti are a distance of more than 22 mm for AU1, AU2, and U points, and a distance of more than 16 mm for the BU point.
Change in vestibular painfulness | 3 months and 6 months
  In cases of vestibular painfulness, light touches with a cotton swab will be performed during the clinical examination on specific points of the vestibular area to determine tender points. The evoked pain will be rated using the Numeric Pain Rating Scale (NPRS), where 0 indicates no pain at all, and 10 indicates the worst imaginable pain. Additionally, the subject will be asked to rate the pain following slow and gentle glowed and lubricated index finger insertion into the vagina to assess the pain intensity associated with finger penetration using the NPRS. The change in pain intensity will be calculated by comparing the initial pain intensity (0-10 points) with the pain intensity after rehabilitation and at follow-up.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Throughout rehabilitation and at 3 months and 6 months
  The rehabilitation team members will monitor treatment-related adverse events throughout the rehabilitation process. Subjects will also be encouraged to report any adverse effects or complications they experience during treatment.
  Adverse events will be classified into five grades based on severity:
  Grade 1 (Mild): Mild adverse events that are asymptomatic or only minimally symptomatic. Grade 2 (Moderate): Moderate adverse events that may cause discomfort but do not significantly interfere with daily activities.
  Grade 3 (Severe): Severe adverse events that are medically significant and may require hospitalization or significant intervention. Grade 4 (Life-threatening): Life-threatening adverse events that pose an immediate risk to life.
  Grade 5 (Death): Adverse events that result in death.
Individual subjects perceptions regarding the helpfulness of the rehabilitation interventions in reducing pelvic floor dysfunction symptoms and enhancing overall functioning | 3 months
  After the rehabilitation, all subjects will be asked to complete a self-reported questionnaire containing close-ended questions, open-ended questions, and global 11-point rating scales (where 0 represents "the specified rehabilitation intervention was not helpful at all," and 10 indicates "maximally helpful"). This questionnaire will assess their individual experiences and attitudes concerning the rehabilitation interventions received and their perceived rehabilitation helpfulness in reducing pelvic floor dysfunctions and functioning impairments.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas, Kauno M. Sav., Lithuania

IPD SHARING:
Plan to Share IPD: No
For now, we do not have enough human and financial resources to share IPD, but if our circumstances change, we are open to reconsidering this decision.